CLINICAL TRIAL: NCT01276301
Title: Relative Bioavailability of BI 10773 Given Alone and Together With Verapamil - an Open-label, Randomised, Crossover Trial in Healthy Subjects
Brief Title: DDI Between BI Empagliflozin (10773) and Verapamil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.43; 2010-023059-27 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — Verapamil; empagliflozin

ARMS (2):
- Reference (Experimental): single dose BI 10773
  Interventions: Drug: BI 10773
- Test (Active Comparator): single dose BI 10773 + single dose verapamil
  Interventions: Drug: Verapamil; Drug: BI 10773

INTERVENTIONS:
Drug: Verapamil — single dose verapamil
  Arms: Test
Drug: BI 10773 — single dose BI 10773
  Arms: Reference
Drug: BI 10773 — single dose BI 10773
  Arms: Test

SUMMARY:
Relative bioavailability of BI 10773 given alone and together with verapamil

ELIGIBILITY:
Inclusion criteria:

healthy male and female subjects

Exclusion criteria:

Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.43.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

REFERENCES:
- [Derived] Macha S, Sennewald R, Rose P, Schoene K, Pinnetti S, Woerle HJ, Broedl UC. Lack of clinically relevant drug-drug interaction between empagliflozin, a sodium glucose cotransporter 2 inhibitor, and verapamil, ramipril, or digoxin in healthy volunteers. Clin Ther. 2013 Mar;35(3):226-35. doi: 10.1016/j.clinthera.2013.02.015. PMID 23497760

RESULTS

PARTICIPANT FLOW:
Groups:
- Empa / Empa Plus Verapamil: A single dose of empagliflozin (empa) 25 mg, followed by a washout period of at least 7 days, followed by a single dose of empagliflozin (empa) 25 mg one hour after administration of a single dose of 120mg verapamil.
- Empa Plus Verapamil / Empa: A single dose of empagliflozin (empa) 25 mg one hour after administration of a single dose of 120mg verapamil, followed by a washout period of at least 7 days, followed by a single dose of empagliflozin (empa) 25 mg.
Period: First Intervention
Arm/Group | Empa / Empa Plus Verapamil | Empa Plus Verapamil / Empa
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Empa / Empa Plus Verapamil | Empa Plus Verapamil / Empa
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Empa / Empa Plus Verapamil | Empa Plus Verapamil / Empa
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: An open label, randomised, two-period crossover trial. The two treatments administered were
  * A single dose of empagliflozin (empa) 25 mg
  * A single dose of empagliflozin (empa) 25 mg one hour after administration of a single dose of 120mg verapamil
  The two treatment periods were separated by a washout period of at least 7 days.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of empagliflozin in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: 0 hours (h), 20 minutes (min), 40min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h and 72h after drug administration
Population: Pharmacokinetic (PK) set: All subjects who had taken at least one dose of trial medication, who had provided at least one observation for at least one primary PK endpoint without an important protocol violation with respect to the PK evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Empa: A single dose of empagliflozin (empa) 25 mg.
- Empa Plus Verapamil: A single dose of empagliflozin (empa) 25 mg one hour after administration of a single dose of 120mg verapamil.
Arm/Group | Empa | Empa Plus Verapamil
Number analyzed (Participants) | 16 | 16
nmol*h/L | 5190 (25.0) | 5340 (25.5)
Statistical Analysis 1: Comparison: Empa vs Empa Plus Verapamil; Ratio calculated as empa plus verapamil divided by empa; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with fixed terms for sequence, period, treatment and random term for subject within sequence; Geometric Mean Ratio = 102.95, 90% CI 2-sided [98.87 to 107.02], Standard Error of Mean 6.5 — Standard error of the mean is actually the Intra-Individual geometric coefficient of variation (gCV)

2. Primary Outcome: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of empagliflozin (empa) in plasma.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol
Arm/Group | Empa | Empa Plus Verapamil
Number analyzed (Participants) | 16 | 16
nmol | 785 (31.5) | 725 (29.1)
Statistical Analysis 1: Comparison: Empa vs Empa Plus Verapamil; Ratio calculated as empa plus verapamil divided by empa; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with fixed terms for sequence, period, treatment and random term for subject within sequence; Geometric Mean Ratio = 92.39, 90% CI 2-sided [85.38 to 99.97], Standard Error of Mean 12.7 — Standard error of the mean is actually the Intra-Individual geometric coefficient of variation (gCV)

3. Secondary Outcome: Area Under the Curve 0 to Time of Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of empagliflozin (empa) in plasma over the time interval from 0 to time of last quantifiable data point.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa | Empa Plus Verapamil
Number analyzed (Participants) | 16 | 16
nmol*h/L | 5140 (25.0) | 5280 (25.7)
Statistical Analysis 1: Comparison: Empa vs Empa Plus Verapamil; Ratio calculated as empa plus verapamil divided by empa; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with fixed terms for sequence, period, treatment and random term for subject within sequence; Geometric Mean Ratio = 102.77, 90% CI 2-sided [98.87 to 106.83], Standard Error of Mean 6.2 — Standard error of the mean is actually the Intra-Individual geometric coefficient of variation (gCV)

4. Secondary Outcome: Time From 0 to Maximum Plasma Concentration (Tmax)
Description: Time from last dosing to the maximum plasma concentration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Empa | Empa Plus Verapamil
Number analyzed (Participants) | 16 | 16
h | 1.50 [1.00 to 2.50] | 1.75 [0.68 to 3.00]

5. Secondary Outcome: Terminal Elimination Rate Constant (λz)
Description: Terminal elimination rate constant in plasma.
  Note: The numbers provide below for standard deviation are of Coefficient of Variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Empa | Empa Plus Verapamil
Number analyzed (Participants) | 16 | 16
1/h | 0.0573 (29.2) | 0.0531 (30.2)

6. Secondary Outcome: Terminal Half-life in Plasma (t1/2)
Description: Terminal half-life of empagliflozin in plasma.
  Note: The numbers provide below for standard deviation are of Coefficient of Variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Empa | Empa Plus Verapamil
Number analyzed (Participants) | 16 | 16
h | 12.1 (29.2) | 13.1 (30.2)

7. Secondary Outcome: Mean Residence Time in the Body After Administration (MRTpo)
Description: Mean residence time of empagliflozin (empa) in the body after oral administration.
  Note: The numbers provide below for standard deviation are of Coefficient of Variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Empa | Empa Plus Verapamil
Number analyzed (Participants) | 16 | 16
h | 9.47 (12.0) | 9.95 (13.8)

8. Secondary Outcome: Apparent Clearance in Plasma After Extravascular Administration (CL/F)
Description: Apparent clearance of empagliflozin (empa) in plasma after extravascular administration.
  Note: The numbers provide below for standard deviation are of Coefficient of Variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Empa | Empa Plus Verapamil
Number analyzed (Participants) | 16 | 16
mL/min | 178 (25.0) | 173 (25.5)

9. Secondary Outcome: Apparent Volume of Distribution Following an Extravascular Dose (Vz/F)
Description: Apparent volume of distribution during the terminal phase following an extravascular dose.
  Note: The numbers provide below for standard deviation are of Coefficient of Variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Empa | Empa Plus Verapamil
Number analyzed (Participants) | 16 | 16
L | 186 (31.8) | 195 (28.8)

10. Other Pre Specified Outcome: Verapamil Plasma Concentration
Description: Verapamil plasma concentration were measured in order to confirm exposure.
  Note: No descriptive statistics was calculated for predose, 49.0 (h) and 73.0 (h), as most of the values were below the limit of quantification (BLQ).
Time Frame: Predose and 1 hour (h), 25h, 49h and 73h after verapamil administration
Population: Treated set (TS) included all subjects who had taken at least one dose of trial medication.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Empa Plus Verapamil
Number analyzed (Participants) | 16
ng/mL
  Planned time: 1.0 (h) | 94.5 (76.3)
  Planned time: 25.0(h) (included 11 participants) | 2.69 (82.2)

11. Secondary Outcome: Clinically Relevant Abnormalities for Physical Examination, Vital Signs, Blood Chemistry and Electrocardiogram (ECG).
Description: Clinically relevant abnormalities for physical examination, vital signs , blood chemistry and Electrocardiogram (ECG). New or abnormal findings were reported as adverse events.
Time Frame: Day1 to Day 11
Population: Treated set (TS) included all subjects who had taken at least one dose of trial medication.
Measure: Number; unit: participants
Arm/Group | Empa | Empa Plus Verapamil
Number analyzed (Participants) | 16 | 16
participants | 0 | 0

12. Secondary Outcome: Assessment of Tolerability by Investigator
Description: Tolerability will be assessed by the investigator according to the categories good, satisfactory, not satisfactory , bad and not assessable.
Time Frame: Within Day 15 to Day 25
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Empa | Empa Plus Verapamil
Number analyzed (Participants) | 16 | 16
percentage of participants
  Good | 100.0 | 87.5
  Satisfactory | 0.0 | 6.3
  Not Satisfactory | 0.0 | 6.3
  Bad | 0.0 | 0.0
  Not assessable | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Day1 to Day 11
Arm/Group | Empa | Empa Plus Verapamil
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 8/16 | 9/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empa (N=16) | Empa Plus Verapamil (N=16)
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Induration (General disorders) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes